CLINICAL TRIAL: NCT06907654
Title: Couples' Affect in Relationships Study
Acronym: Cares
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0357; A171600 (Other: UW Madison); EDUC/COUNSELING PSYCH (Other: UW Madison)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Depression Disorders
Keywords: romantic relationship; long-term relationship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- The Healthy Minds Program (HMP) mobile application (Experimental): Primary participants in the HMP group will be instructed to complete a 4-week intervention through the app.
  Interventions: Device: well-being app
- List of well-being resources (Experimental): Primary participants will be instructed to use a curated list of well-being resources.
  Interventions: Behavioral: List of well-being resources
- Partner - Surveys only (No Intervention): Partner participants will complete surveys their thoughts and feelings.

INTERVENTIONS:
Device: well-being app — The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
  Arms: The Healthy Minds Program (HMP) mobile application
Behavioral: List of well-being resources — Participants will be given a list of resources that promote well-being.
  Arms: List of well-being resources

SUMMARY:
The goal of this clinical trial is to find out whether learning about well-being impacts the thoughts and feelings of romantic couples. The main question it aims to answer is:

* Does gaining knowledge about well-being positively impact individuals and their romantic relationships?

Participants will complete online surveys about their thoughts and feelings.

DETAILED DESCRIPTION:
This study will deliver a meditation-based mobile intervention (The Healthy Minds Program) to one member of a long-term romantic couple and will assess for relationship satisfaction/distress, well-being, and mindfulness in both the primary participant and their partner. The control group will receive a list of well-being-based psychoeducation resources.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Be either married, living together, OR in a dating relationship for at least 12 months
* Proficiency in English
* US citizen or permanent resident
* If non-monogamous, must be able to enroll in the study with a primary partner with whom they spend the majority of their time.
* Use of a smartphone (primary participant only)
* Depression symptoms (≥ 5 on PHQ-9; primary participant only)

Exclusion Criteria:

* Severe physical or sexual relationship aggression during the past 6 months (any item endorsement on 5-item severe IPV screener)
* Endorsement of active suicidality
* History of psychosis or mania
* Prior use of the Healthy Minds Program app
* Prior significant experience with meditation
* Severe hearing impairment that would interfere with the use of an audio-based intervention (primary participant only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Composite of Patient-Reported Outcomes Measurement Information System (PROMIS) Depression | Baseline, Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2-Year Follow-Up
  A measure of feelings of depression scored from 1 to 5 where higher numbers indicate increased feelings of depression. Full range of scores is 28-140.
Change in Second-Person PHQ-9 | Baseline, Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2-Year Follow-Up
  PHQ-9 as assessed by the partner. PHQ-9 is a 9 item survey about how often in the past 2 weeks their partner were bothered by specific problems. It is scored on a 4-point Likert scale, where 0=not at all and 4=nearly every day. Scores range from 0-36, where higher scores indicate more depressive symptoms.
Change in PHQ-9 | Baseline, Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2-Year Follow-Up
  PHQ-9 is a 9 item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale, where 0=not at all and 4=nearly every day. Scores range from 0-36, where higher scores indicate more depressive symptoms.
Change in Couples Satisfaction Index (CSI-16) | Baseline, Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2-Year Follow-Up
  CSI-16 scores can range from 0 to 81. Higher scores indicate higher levels of relationship satisfaction. CSI-16 scores falling below 51.5 suggest notable relationship dissatisfaction.

SECONDARY OUTCOMES:
Change in Sussex-Oxford Compassion for the Self Scale (SOCS-S) | Baseline, Week 4, 3-Month Follow-Up
  SOCS-S is a 20 item survey asking how the participant relates to themself. It is scored on a 5-point Likert scale, where 1 = not at all true and 5 = always true. Scores range from 20-100, with higher scores indicating greater self-compassion.
Relationship Longevity | Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2-Year Follow-Up
  The relationship longevity questionnaire asks participants about their relationship status at the end of study participation.
Change in Problematic and Risky Internet Use Screening Scale (PRIUSS 3) | Baseline, Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2-Year Follow-Up
  PRIUSS 3 is a 3 item questionnaire regarding internet use. It is scored on a 4-point Likert scale where 0=never and 4=very often. Total scores range from 0-12 with higher scores indicating greater problems with internet use.
Change in Second-Person Sussex-Oxford Compassion for the Self Scale (SOCS-S) | Baseline, Week 4, 3-Month Follow-Up
  SOCS-S is a 20 item survey about how your partner might relate to themself. It is scored on a 5-point Likert scale, where 1 = not at all true and 5 = always true. Scores range from 20-100, with higher scores indicating greater self compassion.
Change in Relationship Attribution Measure | Baseline, Week 4, 3-Month Follow-Up
  The relationship attribution measure is a 6 item survey about critical behavior the participant's partner might do. It is scored on a 6-point Likert scale, where 1 = disagree strongly and 6 = agree strongly. Scores range from 6-36, with higher scores indicating greater dissatisfaction with their partner's criticism.
Change in Partner Acceptance Scale | Baseline, Week 4, 3-Month Follow-Up
  The Partner Acceptance Scale is a 5-item scale measuring to what extent the respondent acknowledges his/her partner's imperfections without feeling the urge to change them. It is scored using a 7-point Likert Scale. 1=totally disagree and 7=totally agree. Higher scores indicate greater acceptance of imperfections.
Change in Observed Mindfulness Measure | Baseline, Week 4, 3-Month Follow-Up
  The Observed Mindfulness Measure is a 9 item questionnaire answered by the participant about what they observe about their partner's mindfulness. It is scored on a 5-point Likert scale where 1=not at all and 5=all the time. Scores range from 9-45, with higher scores indicating less mindfulness.
Change in Loneliness Measured by NIH Toolbox Loneliness Score | Baseline, Week 4, 3-Month Follow-Up
  The NIH Toolbox Loneliness is a 5-item questionnaire where participants report how often in the past week they have felt loneliness. It is scored on a 5-point Likert scale where 1 = never to 5 = always. The total possible range of scores is 5-25 where higher scores indicate a greater sense of loneliness.
Change in Anxiety Symptoms Measured by Generalized Anxiety Disorder - 7 (GAD-7) Score | Baseline, Week 4, 3-Month Follow-Up, 1-Year Follow-Up, 2 Year Follow-Up
  The GAD-7 is a 7-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale where 0 = not at all to 3 = nearly every day. The total possible range of scores is 0-21 where higher scores indicate more anxious symptoms.
Change in Healthy Minds (HM) Index | Baseline, Week 4, 3-Month Follow-Up
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the four subscales range as follows: Awareness (0 to 16), Connection (0 to 24), Insight (0 to 12), Purpose (0 to 16) where higher scores indicate more of each quality.
Change in the Mindful Attention Awareness Scale (MAAS) | Baseline, Week 4, 3-Month Follow-Up
  The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place. It is scored on a 6-point Likert scale, where 1=almost always and 6=almost never. Scores range from 15-90 with higher scores indicating lower attention to what is taking place.
Change in Conflict Resolution Scale | Baseline, Week 4, 3-Month Follow-Up
  Conflict Resolution Scale asks participants to select the rating that best describes the outcomes of their disagreements. Scores are summed to get a total score of 0-12 where lower scores indicate worse conflict resolution.
Digital Working Alliance Inventory | Week 4, 3-Month Follow-Up
  The Digital Working Alliance Inventory is a 6-item scale where participants report their working alliance with the HMP app (e.g., "The HMP app supports me to overcome challenges"). It is scored on a 7-point Likert scale where 1 = "strongly disagree" to 7 = "strongly agree." Total scores range from 6 to 42 where higher scores indicate greater working alliance.
Change in Alcohol Use Disorders Identification Test (AUDIT) | Baseline, Week 4, 3-Month Follow-Up
  AUDIT is a 10-item survey asking about the participant's relationship to alcohol. It is scored using various scales depending on the item. Scores range from 0 to 40, with higher scores indicating greater risk for alcohol use disorder.
Change in Cannabis Use Disorders Identification Test - Revised (CUDIT-R) | Baseline, Week 4, 3-Month Follow-Up
  CUDIT-R is an 8-item survey asking about the participant's relationship to cannabis. It is scored using various scales depending on the item. Scores range from 0 to 32, with higher scores indicating greater risk for cannabis use disorder.
Change in Mild-to-moderate IPV Questionnaire | Baseline, Week 4, 3-Month Follow-Up
  Mild-to-moderate IPV Questionnaire is an 7-item survey asking about mild-to-moderate violence in the participant's relationship. It is scored using a 7-point Likert scale, with 0 = never and 6 = more than 20 times. Scores range from 0 to 42, with higher scores indicating greater mild-to-moderate violence in the participant's relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes